CLINICAL TRIAL: NCT05494853
Title: Novel Biomarker Assay for HCC Detection and Monitoring Piedmont Transplant Institute and Genetron Health, Inc.
Brief Title: Novel Biomarker Assay for Biomarker Assay for HCC Detection
Acronym: GTH_HCC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Genetron Health (Industry)
Collaborators: Piedmont Transplant Institute. 1968 Peachtree Road, NW | 77 Building, 6th Floor | Atlanta, GA 30309 (Unknown)
Responsible Party: Sponsor
Other Study IDs: GTH_HCC2022
Record Dates: First submitted 2022-08-08; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Hepato-cellular Carcinoma
Keywords: HCC Screening

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HCC: HCC positive
- Non HCC: HCC negative

SUMMARY:
The primary purpose of this study is to assess the performance feasibility of Genetron's novel HCC liquid biopsy biomarkers assay for early detection. Piedmont Transplant Institute will provide a longitudinally collected blood sample from all HCC cases (mixture of early and advanced stage HCC) and cirrhosis control to Genetron Health after obtaining informed consent.

DETAILED DESCRIPTION:
HCC is a leading cause of cancer-related deaths in the US. Early detection is crucial to improve the outcome of HCC. HCC surveillance is recommended for early detection of HCC in patients with cirrhosis. However, current HCC surveillance tests, such as liver ultrasound and AFP have relatively low accuracy for the detection of early-stage HCC. Genetron Health recently published on novel liquid biopsy biomarker for detection of HCC in China. The biomarker showed excellent performance for the detection of HCC among the at-risk population, most of whom had HBV infection. It is crucial to validate the performance of this novel biomarker in an independent population of patients with different etiology of liver disease outside of China. As this novel biomarker is useful in the detection of small HCC, it may also serve as an excellent biomarker for assessment of treatment response and monitoring of recurrence.

The primary purpose of this study is to assess the performance feasibility of Genetron's novel HCC liquid biopsy biomarkers assay for early detection. Piedmont Transplant Institute will provide a longitudinally collected blood sample from all HCC cases (mixture of early and advanced stage HCC) and cirrhosis control to Genetron Health after obtaining informed consent. Genetron Health will analyze the blood sample and provide data to the PI, for internal review purposes. Should the initial pilot study be successful, the parties will have a discussion to expand the number of cases and control samples and consider conducting a multicenter prospective study.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with HCC (based on histology or radiology according to AASLD guideline) or liver cirrhosis (based on the clinical history of hepatic encephalopathy, thrombocytopenia, radiologic features of the nodular liver, features of portal hypertension such as ascites, splenomegaly, or MR elastogram or fibroscan showing result consistent with cirrhosis)
* Willing and able to provide informed consent to participate in this study

Exclusion Criteria:

* Unable to provide blood samples
* Age less than 18 years of age
* Patient who have active cancers (excluding HCC) in the past five years, except for nonmelanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cirrhotic patients without HCC, early intermediate stage HCC, advanced-stage HCC, and patients who remained in remission after curative treatment. ASH, fatty liver, NASH, HCV are the most common etiology of HCC and cirrhosis in our cohort.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
HCC screening positive | 2 years
  Data will suggest the probability of HCC

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Qu C, Wang Y, Wang P, Chen K, Wang M, Zeng H, Lu J, Song Q, Diplas BH, Tan D, Fan C, Guo Q, Zhu Z, Yin H, Jiang L, Chen X, Zhao H, He H, Wang Y, Li G, Bi X, Zhao X, Chen T, Tang H, Lv C, Wang D, Chen W, Zhou J, Zhao H, Cai J, Wang X, Wang S, Yan H, Zeng YX, Cavenee WK, Jiao Y. Detection of early-stage hepatocellular carcinoma in asymptomatic HBsAg-seropositive individuals by liquid biopsy. Proc Natl Acad Sci U S A. 2019 Mar 26;116(13):6308-6312. doi: 10.1073/pnas.1819799116. Epub 2019 Mar 11. PMID 30858324